CLINICAL TRIAL: NCT01104285
Title: Chest Tube Drainage of Transudative Pleural Effusions Hastens Liberation From Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Sidney Tessler, Director, Pulmonary and Critical Care Medicine, Maimonides Medical Center
Other Study IDs: 10/03/VA02
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Results first posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-04

CONDITIONS: Liberation From Mechanical Ventilation

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard care: Treatment of pleural effusion with diuresis
- Chest tube: Treatment of pleural effusion with diuresis and chest tube

SUMMARY:
The purpose of this study is to determine whether chest tubes to drain transudative pleural effusions helps patients come off mechanical ventilation earlier.

ELIGIBILITY:
Inclusion Criteria:

* Patients with transudative pleural effusion and requiring mechanical ventilation

Exclusion Criteria:

* Patients with coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 112 patients standard; 86 patients chest tube
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yizhak Kupfer, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Derived] Kupfer Y, Seneviratne C, Chawla K, Ramachandran K, Tessler S. Chest tube drainage of transudative pleural effusions hastens liberation from mechanical ventilation. Chest. 2011 Mar;139(3):519-523. doi: 10.1378/chest.10-1012. Epub 2010 Aug 5. PMID 20688921 (Retraction: PMID 22215847 Chest. 2012 Jan;141(1):284)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | Chest Tube
Started | 112 | 86
Completed | 112 | 86
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Chest Tube | Total
Number analyzed (Participants) | 112 | 86 | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 10 | 27
  >=65 years | 95 | 76 | 171
Age Continuous [Mean (Standard Deviation); unit: years] | 78 (9) | 77 (11) | 78 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 53 | 124
  Male | 41 | 33 | 74
Region of Enrollment [Number; unit: participants]
  United States | 112 | 86 | 198

OUTCOME MEASURES:

1. Primary Outcome: Total Days of Mechanical Ventilatory Support
Time Frame: days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Care | Chest Tube
Number analyzed (Participants) | 112 | 86
days | 6.51 (1.5) | 4.02 (3.9)

ADVERSE EVENTS:
Arm/Group | Standard Care | Chest Tube
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/86
Other Adverse Events (participants affected / at risk) | 0/112 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes